CLINICAL TRIAL: NCT04537754
Title: Clinical Comparison of LED- and Diode Laser-activated Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aybuke Uslu, specialist of restorative dentistry, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AUslu
Record Dates: First submitted 2020-07-08; First posted 2020-09-03 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Color; Change Teeth, Posteruptive
Keywords: In-office tooth bleaching; Diode laser; LED; color change; tooth-sensitivity; temperature
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- clinician (Experimental): Comparison of LED and diode laser
  Interventions: Device: bleaching device

INTERVENTIONS:
Device: bleaching device — activated bleaching
  Other Names: whitness hp, FGM; Radii plus LED,SDI; Epic X, Biolase

SUMMARY:
To clinically compare the effects of LED- or Diode laser-activated bleaching on colour change, tooth-sensitivity, gingival-irritation and temperature variation over 9-months.

Thirty-five patients with tooth colour A2 or higher will be included in the study. In a split-mouth design, using a 35% HP bleaching agent (Whiteness HP); one side of each mouth will be randomly activated by a diode laser (Epic X) and the other side by an LED (Radii Plus) light-source. During bleaching, the temperature variations will be recorded using a thermocouple from the buccal surface of canine teeth. Colour change (ΔSGU, ΔE) will be evaluated by subjective (Vita classic/bleached guide) and objective methods (spectrophotometry) before treatment and immediately, 48h, 1 week, 1, 6, 9 months after. Tooth-sensitivity and gingival- irritation will be assessed by visual analogue scale (VAS) and Gingival Index.

DETAILED DESCRIPTION:
Objective: The aim of this split-mouth, randomized clinical study is to evaluate the effect of LED or Diode laser-activated bleaching applications on colour change, tooth sensitivity, gingival irritation and temperature variation with 35% hydrogen peroxide bleaching gel after 9 months. Material and Methods: Thirty-five patients with anterior teeth without caries and no restoration will be included in this study. In a split-mouth design, a bleaching agent containing 35% HP (Whiteness HP, FGM) will be used, one side of each jaw will be activated by a diode laser (Epic X, Biolase) and the other side will be activated by an LED (Radii Plus, SDI) light source. During the bleaching treatments, the temperature variations will be recorded using a thermocouple (DT-3891G K type Thermometer datalogger, CEM Instruments) from the buccal surface of canine teeth. Tooth sensitivity will be assessed by Visual Analogue Scale (VAS) before the treatment and during, immediately, 48 hours, 1 week, 1, 6 and 9 months after. Color change will be evaluated by subjective (Vita Classic and Vita 3D Master Bleachguide) and objective methods (Vita Easy Shade, spectrophotometer) before the treatment and immediately, 48 hours, 1 week, 1, 6 and 9 months after. Color change (ΔE and ΔSGU) will be performed by analysis of variance in repeated measurements. Multiple comparisons will be evaluated by Bonferroni test. Temperature variation will be evaluated by t-test in dependent groups. Tooth sensitivity will be analyzed using Friedman test. Wilcoxon test will be used to compare two light sources (Diode Laser/ LED) in each time period (p< 0.05).

ELIGIBILITY:
Inclusion Criteria:

* healthy vital anterior teeth without restorations which have A2 or darker tooth shade on Vita Classical Scale (Vita Classical Scale, VITA Zahnfabrik, Bad Säckingen, Germany).

Exclusion Criteria:

* Pregnant or lactating woman smokers Participants with periodontal diseases, tooth sensitivity internal tooth discoloration (tetracycline/ fluorosis stains), exposed engine, peroxides allergy malpositioned teeth

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Colour change | Baseline (before the treatment) and 48 hours, 1 week, 1, 6 and 9 months after.
  Colour change will be evaluated by subjective (Vita Classic and Vita 3D Master Bleachguide) and objective methods (Vita Easy Shade, spectrophotometer).
temperature | Procedure (During the bleaching treatments)
  During the bleaching treatments, the temperature variations will be recorded using a thermocouple (DT-3891G K type Thermometer datalogger, CEM Instruments) from the buccal surface of canine teeth.
Tooth sensitivity | Baseline (before the treatment) and 48 hours, 1 week, 1, 6 and 9 months after.
  Tooth sensitivity will be assessed by Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: A. Ruya Yazici, Prof., Study Director — Hacettepe University
Locations (1):
- Aybuke Uslu, Ankara, Turkey (Türkiye)